CLINICAL TRIAL: NCT02523638
Title: An Open-label, Single Arm, Phase III Study to Assess the Self-administration of AOP2014 Using a Pre-filled Pen, Developed for the Treatment of Polycythemia Vera Patients
Brief Title: Study to Assess the Self-administration of AOP2014 Using a Pen, Developed for the Treatment of Polycythemia Vera Patients
Acronym: PEN-PV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Collaborators: PharmaEssentia Corporation (Co-Sponsor for USA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEN-PV; 2014-001356-31 (EudraCT Number)
Record Dates: First submitted 2015-06-12; First posted 2015-08-14 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Polycythemia Vera
Keywords: Pegylated-Proline-interferon alpha-2b (AOP2014); Polycythemia Vera; PEN-PV; PROUD-PV; CONTINUATION-PV; AOP Orphan; Polycythemia; Hematologic Diseases; Myeloproliferative Disorders; Bone Marrow Diseases; Interferon-alpha; Peginterferon alfa-2b
MeSH Terms: conditions — Polycythemia Vera; Polycythemia; Hematologic Diseases; Myeloproliferative Disorders; Bone Marrow Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pegylated- Proline-Interferon alpha-2b (Other): Pegylated-Proline-Interferon alpha-2b in a Pre-filled Pen single arm
  Interventions: Drug: Pegylated-Proline-Interferon alpha-2b in a Pre-filled Pen

INTERVENTIONS:
Drug: Pegylated-Proline-Interferon alpha-2b in a Pre-filled Pen — Subjects will continue to receive the dosage which delivers the optimal disease response (hematocrit [Hct]<45%, platelets [PLTs]<400 x 109/L and leukocytes [WBCs]<10 x 109/L), as determined in the PROUD-PV study, preferably at the level of target blood values.
  Other Names: AOP2014

SUMMARY:
Polycythemia Vera (PV) is a disease of bone marrow stem cells that manifests in a drastic increase of red blood cells and frequently also of white blood cells. The "thickening" of the blood in relation with a modified function of the cells has several consequences like increased blood pressure, pruritus of the skin, fatigue, disturbed blood circulation in the brain as well as fingers and toes and an increased risk of arterial and venous thrombosis (thrombosis is the formation of a blood clot in a vessel); like stroke, cardiac infarction, deep vein thrombosis in the legs. In case of a strong increase of platelets there is an additional risk of bleedings. As the disease progresses the size of spleen and liver increased in most cases and the bone marrow shows signs of fibrosis. In some cases of PV a progression at a later time point to a leukemia (increased formation of white blood cells) can occur.

The aim of this study is to assess the ease of AOP2014 self-administration using dedicated questionnaires.

* To assess safety and tolerability: adverse events (AEs), laboratory parameters, electrocardiogram (ECG) throughout study.
* To assess maintenance of the blood efficacy parameters Hct (Hematocrit), WBC (white blood cells) and PLTs (platelets) and spleen size (comparing values at Visit P7 vs. values at Visit P1).
* To assess the feasibility of AOP2014 self-administration: defined as the ability of the patients to use the pen as a self-administration tool (ease of handling, safety, tolerability and efficacy).

DETAILED DESCRIPTION:
This is a Phase III, single-arm study performed in patients who completed the AOP2014 arm of the PROUD-PV study or are currently participating in the CONTINUATION-PV study. After signing the informed consent form (ICF), approximately 30 patients will be enrolled consecutively into the study at participating sites according to the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who either completed the 12 months AOP2014 treatment arm of the PROUD-PV study, or are currently participating in the CONTINUATION-PV, and at the "EoT visit" (End of treatment visit) of the PROUD-PV study or two weeks after the last assessment visit of the CONTINUATION-PV study, fulfill at least one of the following criteria:

   * Normalization of at least two out of three main blood parameters (Hct (Hematocrit), PLTs (Platelets) and WBCs (white blood cells) if these parameters were moderately increased (Hct<50%, WBCs<20 x 109/L, PLTs<600 x 109/L) at baseline visit of the PROUD-PV study, OR
   * >35% decrease of at least two out of three main blood parameters (Hct, PLTs and WBCs) if these parameters were massively increased (Hct>50%, WBCs>20 x 109/L, PLTs >600 x 109/L), at baseline visit of the PROUD-PV study, OR
   * Normalization of spleen size, if spleen was enlarged at baseline visit of the PROUD-PV study, OR
   * Otherwise a clear, medically verified benefit from treatment with AOP2014 (e.g. normalization of disease-related micro-vasculatory symptoms, substantial decrease of JAK2 (Januskinase 2) allelic burden).
2. Signed written ICF.

Exclusion Criteria:

Withdrawal criteria, as specified in the PROUD-PV and CONTINUATION-PV studies, which mandate treatment discontinuation.

1. Non-recovery from the AOP2014 related toxicities to the grade (usually, Grade I) which allows continuation of the treatment.
2. HADS (Hospital Anxiety and Depression Scale) score of 11 or higher on either or both of the subscales, and /or development or worsening of clinically significant depression or suicidal thoughts.
3. Progressive and clinically significant increase of liver enzyme levels despite dose reduction, or if such increase is accompanied by increased bilirubin level, any signs or symptoms of a clinically significant autoimmune disease.
4. Clinically significant development of a new ophthalmologic disorder, or worsening of a pre-existing one, during the study.
5. Loss of efficacy of AOP2014 or any comparable situation where no further benefits of treatment continuation are expected by the investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To evaluate ease of self-administration of AOP2014 | 3 months
  To evaluate ease of self-administration of AOP2014 as assessed by staff and patients using dedicated questionnaires, using rates of full success and failure rates (defined in the statistics section of the synopsis).

SECONDARY OUTCOMES:
Adverse Event | 3 month
  biweekly, using dedicated questionnaires
number of phlebotomies | 3 months
  biweekly
Disease response | 3 months
  The main efficacy evaluation criterion will be disease response defined as:
  • Hct (Hematocrit)< 45% without phlebotomy (at least 3 months since the last phlebotomy).
  The hematological parameters will be measured by the local laboratories at clinical sites.
Disease response | 3 months
  The main efficacy evaluation criterion will be disease response defined as:
  • PLTs (Platelets)< 400 x 109/L. The hematological parameters will be measured by the local laboratories at clinical sites.
Disease response | 3 months
  The main efficacy evaluation criterion will be disease response defined as:
  • WBCs (White blood cells)< 10 x 109/L. The hematological parameters will be measured by the local laboratories at clinical sites.
blood parameters | 3 months
  first biweekly than monthly
  The main efficacy evaluation criterion will be disease response defined as:
  • Hct< 45% without phlebotomy (at least 3 months since the last phlebotomy). The hematological parameters will be measured by the local laboratories at clinical sites.
blood parameters | 3 months
  first biweekly than monthly
  The main efficacy evaluation criterion will be disease response defined as:
  • WBCs< 10 x 109/L. The hematological parameters will be measured by the local laboratories at clinical sites.
blood parameters | 3 months
  first biweekly than monthly
  The main efficacy evaluation criterion will be disease response defined as:
  • PLTs< 400 x 109/L. The hematological parameters will be measured by the local laboratories at clinical sites.
spleen size | 3 months
  locally, Sonography will be used for measuring the spleen size (length). at Visit 1 and at the End of the study (week 12)
disease related symptoms | 3 months
  biweekly, using dedicated questionnaires
protocol-specific adverse events of special interest | 3 months
  biweekly, using dedicated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Gisslinger, MD, Principal Investigator — Med Uni Wien
Locations (35):
- Austria (7):
  - LKH Graz, Graz
  - University Hospital Innsbruck, Innsbruck
  - Elisabethinen Hospital Linz, Linz
  - Salzburg Regional Hospital, Salzburg
  - Hanusch Hospital, Vienna
  - Medical University Vienna, Vienna
  - Hospital Wels-Grieskirchen, Wels
- Bulgaria (2):
  - Specialized Hospital for Active Treatment of Hematological Diseases, Sofia
  - Multiprofile Hospital for Active Treatment - Hristo Botev, Vratsa, First Department of Internal Medicine, Vratsa
- Czechia (5):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - Institute of Hematology and Blood Transfusion, Prague
  - University Hospital Kralovske Vinohrady, Prague
  - University Hospital Motol, Prague
- France (3):
  - Institute Paoli-Calmettes, Marseille
  - Hospital Saint-Louis, Paris
  - Clinical Research Center CIC, Poitiers
- Hungary (5):
  - St Istvan and St Laszlo Hospital of Budapest, Budapest
  - University of Debrecen, Debrecen
  - Bekes County Pandy Kalman Hospital, 1st Department of Medicine, Hematology, Gyula
  - Kaposi Mor County Teaching Hospital, Kaposvár
  - University of Szeged, Albert Szent-Gyorgyi Clinical Center, Koranyi fasor 6, Szeged
- Poland (6):
  - Andrzej Mielecki Independent Public Clinical Hospital of Medical University of Silesia in Katowice, Katowice
  - University Hospital in Cracow, Krakow
  - Independent Public Teaching Hospital No.1 in Lublin, Lublin
  - Fryderyk Chopin Provincial Specialized Hospital, Rzeszów
  - Nicolaus Copernicus Municipal Specialist Hospital, Torun
  - Institute of Hematology and Transfusion Medicine, Warsaw
- Slovakia (2):
  - University Hospital with Outpatient Clinic F.D. Roosevelt, Banská Bystrica
  - Saint Cyril and Metod University Hospital Bratislava, Bratislava
- Ukraine (5):
  - Cherkasy Regional Oncology Center, Regional Treatment and Diagnostics Hematology Center, Cherkasy
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Dnipropetrovsk
  - National Research Center for Radiation Medicine, Institute of Clinical Radiology, Kiev
  - Institute of Blood Pathology and Transfusion Medicine, Lviv
  - O.F. Herbachevskyi Regional Clinical Hospital, Zhytomyr